CLINICAL TRIAL: NCT02659033
Title: Impact of the Choice of 3rd Generation Cephalosporins on the Emergence of Resistance in the Microbiota Intestinal.
Acronym: CEREMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC13-179 / P140904; 2014-005485-30 (EudraCT Number)
Record Dates: First submitted 2016-01-05; First posted 2016-01-20 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Emergence of Bacterial Resistance to Antibiotics
Keywords: microbiota; resistant bacteria
MeSH Terms: interventions — Ceftriaxone; Third Generation Cephalosporins; Cefotaxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ceftriaxone (Active Comparator): healthy volunteer who receive ceftriaxone
  Interventions: Drug: ceftriaxone
- cefotaxime (Active Comparator): healthy volunteer who receive cefotaxime
  Interventions: Drug: Cefotaxime

INTERVENTIONS:
Drug: ceftriaxone — ceftriaxone (1 gram per day)
  Other Names: cephalosporin 3rd generation
  Arms: ceftriaxone
Drug: Cefotaxime — cefotaxime (1 gram every 8 hours)
  Other Names: cephalosporin 3rd generation
  Arms: cefotaxime

SUMMARY:
CEREMI is an open, randomised prospective study in parallel groups in healthy volunteers. This study compare the effect of a monotherapy by ceftriaxone or cefotaxime on the emergence of resistance of enterobacteria to 3rd-generation cephalosporins within the intestinal microbiota. Each volunteer will be treated for 3 days by either ceftriaxone (1 gram per day) or cefotaxime (1 gram every 8 hours).

DETAILED DESCRIPTION:
Selection of resistant bacteria within the microbiota constitutes the main mechanism for the emergence and the diffusion of bacterial resistance to antibiotics. Ceftriaxone is a 3rd generation cephalosporin that exposes the intestinal microbiota to an important selecting pressure, due to its high biliary clearance. It is thereby suspected to have an important role in the emergence of resistance of enterobacteria to 3rd generation cephalosporins. Its pharmacokinetics features allow a once daily administration, and it is more largely used than cefotaxime, which requires ter in die injections but whose mainly urinary elimination suggest a lower impact on the intestinal microbiota.

Our hypothesis is that ceftriaxone exerts a higher selecting pressure on the intestinal microbiota than cefotaxime.

Our main objective is to compare the effect of a monotherapy by ceftriaxone or cefotaxime on the emergence of resistance of enterobacteria to 3rd-generation cephalosporins within the intestinal microbiota.

Secondary objectives include :

* Comparison of the effect of ceftriaxone and cefotaxime on the counts of (i) total enterobacteria, (ii) 3rd generation cephalosporins resistant enterobacteria according to the resistance mechanism, (iii) colonisation resistance in the intestinal microbiota
* Pharmacokinetic analysis of cefotaxime and ceftriaxone at steady-state, and link between plasma and fecal expositions to each antimicrobial
* Analysis of the association between individual exposition to ceftriaxone and cefotaxime and their impact on the intestinal microbiota.

The main evaluation criteria is the area under the curve of the 3rd generation cephalosporins resistant enterobacteria in the intestinal microbiota between D0 and D7.

Secondary evaluation criteria include :

* Bacterial and fungal AUC (area under the curve) in the intestinal microbiota between D0 and D7 and between D0 and D15. Proportion of patients with 3rd generation cephalosporins resistant enterobacteria and proportion of patients with non commensal bacteria and fungi in the intestinal microbiota at D30, at D90 and at D180.
* Studied pharmacokinetic parameters : total bocy clearance, volume of distribution, half life. Studied plasma exposition parameters : AUC, maximal and minimal concentration at steady-state. Studied fecal exposition parameter : AUC between D0 and D7.
* Association between plasma and fecal exposure and AUC of bacterial and fungal counts between D0 and D7.

Methodology :

Open, randomised prospective study in parallel groups in healthy volunteers. Each volunteer will be treated for 3 days by either ceftriaxone (1 gram per day) or cefotaxime (1 gram every 8 hours). Fecal samples will be collected before (3 samples, D-14, D-7 and D-1) and after the first administration of the antibiotic (D1, D2, D3, D4, D7, D10, D15, D30, D90, D180).

Bacterial analysis of the fecal samples will be performed blindly from the treatment group. Drug plasma concentration will be determined at steady-state (T0, T0.5h, T1h, T2h, T4, T6h for cefotaxime and T0, T0.5h, T1h, T2h, T4, T8h for ceftriaxone). Drug concentration in the feces will be measured on the samples obtained between D0 and D7.

Pharmacokinetic analysis will be performed using the population approach. All statistical analysis will be performed using non parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Volunteer regarded as healthy after detailed examination
* Subject whose entourage (person living under the same roof) does not present any chronic disease throughout the course and did not receive antibiotics within 15 days.
* Effective contraception for women in reproductive age and negative pregnancy test before inclusion
* Normal intestinal passage (one stool per day)
* Negative urinalysis for toxic substances
* Normal blood test (including blood and platelets counts, prothrombin, ionograms, Liver function tests)
* Negative HIV and HCV (hepatitis C virus) test, no HBV (hepatitis B virus)chronic infection
* Normal weight (BMI comprised between 19 and 29 kg/m²)
* Freely obtained consent
* Health insurance beneficiary

Exclusion Criteria:

* Antibiotic therapy in the previous 6 months
* Hospitalisation in the previous 12 months;
* Active infection
* Ongoing treatment
* Any chronic disease
* Allergy to one of the study drugs
* Any contraindications to β-lactam therapy in particular to penicillins or cephalosporins
* Pregnancy or no effective contraception, suckling women
* Subject, as determined by the investigating physician, could not observing during the study, or unable to communicate because of language or mental disorders barrier;
* Subject participating simultaneously in another biomedical research
* Subject can not be contacted in case of emergency;
* Subject about legally protected under tutorship or curators;
* Subject deprived of freedom under judicial or administrative constraints

Secondary exclusion criteria

* No pre-treatment stool sample obtained
* More than one stool sample missing from D1 to D7

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03; Primary Completion 2016-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The area under the curve of the 3rd generation cephalosporins resistant enterobacteria in the intestinal microbiota between D0 and D7. | within the first 7 days

SECONDARY OUTCOMES:
The area under the curve of enterobacteriaceae resistant to C3G accounts (regardless of the resistance mechanism) from D0 to D15 in each treatment group. | within the first 15 days
Proportion of patients with 3rd generation cephalosporins resistant enterobacteria in the intestinal microbiota (regardless of the resistance mechanism) at D30 at D90 and at D180 in each treatment group. | D30, D90 and D180
Area under the curve of enterobacteriaceae resistant to C3G accounts distinguishing the resistance mechanism (B lactamase,plasmid cephalosporinase or cephalosporinase) from D0 to D15 in each treatment group. | within the first 15 days
Proportion of patients with 3rd generation cephalosporins resistant enterobacteria in the intestinal microbiota (distinguishing the resistance mechanism) at D30 at D90 and at D180 in each treatment group. | D30, D90 and D180
Area under the curve of total coliform accounts from D0 to D 7 and D0 to D15 in each treatment group. | within the first 15 days
Change in total coliform accounts between D0 and D30 between D0 and D90 and between D0 and D180 in each treatment group. | D30, D90 and D180
The area under the curve of aeruginosa accounts, S. aureus, Enterococcus spp., Clostridium difficile and yeasts from D0 to D7 and D0 to D15 in each treatment group. | within the first 15 days
The area under the curve of β-lactamase activity of the intestinal microbiota from D0 to D7 and D0 to D15 in each treatment group. | within the first 15 days
Proportion of patients with β-lactamase activity in the stools at D30, D90 and D180 in each treatment group. | D30, D90 and D 180

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Duval, Profesor, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Burdet C, Grall N, Linard M, Bridier-Nahmias A, Benhayoun M, Bourabha K, Magnan M, Clermont O, d'Humieres C, Tenaillon O, Denamur E, Massias L, Tubiana S, Alavoine L, Andremont A, Mentre F, Duval X; CEREMI Group. Ceftriaxone and Cefotaxime Have Similar Effects on the Intestinal Microbiota in Human Volunteers Treated by Standard-Dose Regimens. Antimicrob Agents Chemother. 2019 May 24;63(6):e02244-18. doi: 10.1128/AAC.02244-18. Print 2019 Jun. PMID 30936104